CLINICAL TRIAL: NCT00703040
Title: HIV-Related Care Engagement: Linkage to Care and Care-Seeking for HIV-Infected Adolescents, Phase I
Brief Title: Linkage to Care - Part I
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 066a
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-02

CONDITIONS: HIV
Keywords: Care engagement; Linkage to care; HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Component 1: Existing linkage to care protocols will be obtained from the 15 sites. This component does not involve study subjects.
- Component 2: Person-to-person or telephone interviews with ATN clinical site staff and staff from their community partners will be audio-taped.
- Component 3: Notes from direct observation of the linkage to medical care process within sites will be taken.

SUMMARY:
This first phase of a two-phase study involves three components:

1. Review of existing linkage-to-care protocols and sources of referrals for care;
2. Semi-structured telephone or face-to-face interviews with a minimum of two personnel per site who are associated with linkage to medical care. (Preference will be given to personnel with direct experience in linkage to care); and
3. Structured observations of referral sessions.

ELIGIBILITY:
Inclusion Criteria:

* Component 1: Documents identified by clinical site personnel as pertaining to post-test counseling, linkage to care, or standard operating procedures addressing post-test counseling and linkage to care.
* Component 2: Persons employed by one of the AMTUs or an identified linkage-to-care partner and work as clinical staff or a case-manager or is a person familiar to linkage to care; or persons involved in posttest counseling and linkage-to-care processes. Clinical staff and case managers are chosen based on direct experience in the assistance of HIV seropositive youth obtaining medical care. This definition includes, but is not limited to, physicians, nurses, psychologists, social workers, and case managers (who may have diverse professional backgrounds).
* Component 3: All AMTU sites will be included.

Exclusion Criteria:

* Component 1: No a priori exclusions.
* Component 2: No a priori exclusions.
* Component 3: No a priori exclusions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Component 1: The object of study is a collection of documents on existing linkage-to-care protocols and does not constitute a population. Component 2: Ideally, a minimum of two clinical staff and/or case managers from each of 15 AMTU and a minimum of one staff member representing the AMTU's community partners/sites where linkage to care activities occur. Component 3- Structured Observations: Clinical site staff providing linkage to care counseling. Please note that patients are not part of this study population. See Section 5.3 and Section 10.0 for additional details.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2008-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Describe and evaluate community screening standards and practices. | 1 year
Describe and evaluate the relationships of screening venues with care-providing venues. | 1 year
Describe and evaluate referral and intake protocols. | 1 year
Describe and evaluate care adherence support (including support from both clinical and non-clinical sources). | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: J. Dennis Fortenberry, MD, Study Chair — Adolescent Trials Network
Locations (7):
- United States (7):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Childrens Diagnostic&Treatment Center, Fort Lauderdale, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Mount Sinai Medical Center, Manhattan, New York
  - Montefiore Medical Center, The Bronx, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Childrens Research Hospital, Memphis, Tennessee

REFERENCES:
- See also: Adolescent Trials Network website — http://www.atnonline.org